CLINICAL TRIAL: NCT01413438
Title: Prospective, Randomized Controlled Trial of Surgical Resection Prior to Bevacizumab Therapy for Recurrent Glioblastoma Multiforme
Brief Title: Bevacizumab With or Without Surgery for Adult Glioblastomas
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110204; 11-N-0204
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2013-09-26

CONDITIONS: Glioblastoma; Brain Neoplasm
Keywords: Bevacizumab; Quality of Life; Glioblastoma Multiforme; Neurosurgery; Glioblastoma; GBM; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Craniotomy

INTERVENTIONS:
Procedure: Craniotomy

SUMMARY:
Background:

- Glioblastoma (GBM) is the most common malignant brain tumor in adults. Patients with GBM are usually treated with surgery, radiation, and chemotherapy. Despite this treatment, most GBMs start growing again. Bevacizumab, a chemotherapy drug, has shown promise in slowing the growth of GBMs. More research is needed to find out whether having surgery before starting bevacizumab is more effective than bevacizumab alone.

Objectives:

- To compare surgery plus bevacizumab to bevacizumab alone in adults with glioblastoma.

Eligibility:

- Individuals at least 18 years old whose glioblastoma has come back after treatment.

Design:

* All participants will be screened with a physical exam, medical history, blood tests, and imaging studies.
* Participants will be divided into two groups. One group will have surgery followed by bevacizumab. The other group will have the drug without surgery.
* The first group will have surgery as soon as possible and will begin bevacizumab 4 weeks after surgery. The second group will start the drug as soon as possible.
* Both groups will receive the drug as an infusion every 2 weeks. They will be monitored with frequent blood tests and imaging studies. The infusions will continue for as long as the drug is effective at preventing tumor regrowth.
* Participants will be contacted every 4 weeks after they stop taking bevacizumab. They will answer followup questions either in person or by telephone.

DETAILED DESCRIPTION:
Objective

The objective of this prospective randomized controlled study is to determine the overall survival benefit of tumor resection in patients with recurrent glioblastoma multiforme (GBM).

Study Population

This study will recruit 42 adults with a diagnosis of recurrent grade 4 astrocytoma into each of two arms, for a total of 84 patients. All participants will be good candidates for elective surgical resection of their tumors according to the previously established NIH Recurrent Glioma Scale (NRGS), which uses performance status, tumor volume, and tumor involvement of critical/eloquent brain areas as prognostic criteria. Patients who require biopsy only or have previously been treated with bevacizumab will be excluded.

Design

Participants will be stratified by NRGS score (NRGS 0 or NRGS 1-2) and randomized to surgery followed by bevacizumab or to bevacizumab alone. Patients assigned to the surgical arm will undergo their procedure within 28 days of randomization. Treatment with bevacizumab at a dose of 10 mg/kg every 2 weeks will begin at least 28 days later to allow adequate craniotomy wound healing. Patients assigned to the non-surgical arm will start bevacizumab at a dose of 10 mg/kg every 2 weeks immediately. MRI evaluations will take place within 72 hours of surgery to assess extent of resection, 28 days postoperatively, 96 hours after starting bevacizumab, and then every 28 days until tumor progression is documented. Follow-up assessments will take place every 28 days while on bevacizumab until tumor progression. Once progression is established, patients will be free to pursue further surgical and/or medical salvage therapy as they wish. Patients will be followed until their time of death.

Outcome Measures

The primary outcome measure is median overall survival from the date bevacizumab is started. Secondary outcome measures include the rate of progression-free survival 6 months after starting bevacizumab, median progression-free survival, overall survival rates at 6 and 12 months after starting bevacizumab, objective response rate, health-related quality of life, change in KPS of 20 points or more, time to need for additional tumor therapy, and use of corticosteroids.

ELIGIBILITY:
* INCLUSION CRITERIA:

Previous diagnosis of supratentorial GBM established by WHO histological criteria

Age 18 or older

NRGS score of 0 to 2 established by the following criteria:

* KPS 80 or less (1 point)
* Tumor volume 50 cc or greater (1 point)
* Tumor involvement of at least 2 of the following brain areas (1 point):

  * Motor cortex
  * Language cortex
  * Areas directly adjacent to the proximal (M1 and/or M2) middle cerebral artery

Received initial treatment for GBM with:

* External beam radiation therapy
* Nitrosourea or temozolomide chemotherapy
* Biopsy, subtotal or gross total resection

Evidence of recurrence, defined as the appearance or enlargement since previous imaging of a contrast-enhancing mass on T1-weighted MRI

Have a non-deep (involving basal ganglia, thalamus, or periventricular region), non-diffuse recurrence judged to be resectable by a neurosurgeon

Able to provide informed consent

EXCLUSION CRITERIA:

NRGS score of 3

Patients requiring biopsy only or other procedures where the goal is not tumor cytoreduction

Patients who require urgent or emergency surgery due to symptoms of raised intracranial pressure or herniation

Patients who have already received bevacizumab therapy

Contraindication to surgery as determined by a neurosurgeon, including bleeding diathesis, unacceptable pulmonary or cardiovascular risk, significant wound healing concerns, or tumor recurrence judged to be inoperable, inaccessible, or diffuse

Contraindication to bevacizumab as determined by a neuro-oncologist, including unacceptable end organ function, evidence of acute intracranial hemorrhage, or recent or active use of anticoagulants

Contraindication to MRI scanning as determined by a radiologist, including pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, or shrapnel fragments

Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07-15; Primary Completion 2013-09-26 (Actual); Study Completion 2013-09-26 (Actual)

PRIMARY OUTCOMES:
Median Overall Survival | 2 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) at 6 months & median PFS in each arm, objective response rate by the RANO criteria (OR), and overall survival rate at 6 and 12 months in each arm, compare rate of change in health-related quality of life. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John K Park, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)

REFERENCES:
- [Background] Arko L, Katsyv I, Park GE, Luan WP, Park JK. Experimental approaches for the treatment of malignant gliomas. Pharmacol Ther. 2010 Oct;128(1):1-36. doi: 10.1016/j.pharmthera.2010.04.015. Epub 2010 Jun 8. PMID 20546782
- [Background] Clarke J, Butowski N, Chang S. Recent advances in therapy for glioblastoma. Arch Neurol. 2010 Mar;67(3):279-83. doi: 10.1001/archneurol.2010.5. PMID 20212224
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009